CLINICAL TRIAL: NCT07326839
Title: Optimization of Blood Uric Acid Control in Obese Gout Patients by Orlistat-Mediated Metabolic Remodeling and Intensive Weight Management: A Randomized Controlled Trial
Brief Title: Orlistat and Weight Management for Uric Acid Control in Obese Gout: A RCT
Acronym: OWMUAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XueMei Guo (Other)
Collaborators: Shengjing Hospital (Other); The People's Hospital of Liaoning Province (Other)
Responsible Party: Sponsor-Investigator, XueMei Guo, General Hospital of Shenyang Military Region, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025JH2/101800052
Record Dates: First submitted 2025-12-19; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Gout; Obesity
Keywords: Obese; Gout; Orlistat; Metabolic Reprogramming; Weight Control; Uric acid; AMPK; HIF1; NLRP3
MeSH Terms: conditions — Gout; Obesity | interventions — Orlistat; Febuxostat

STUDY DESIGN:
Intervention Model Description: Randomized open-label, two-arm parallel control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental Group (Experimental): The experimental Group received orlistat 120mg tid+ standard ULT (e.g., febuxostat 40mg qd) + basic lifestyle advice (low-purine diet and exercise guidance).
  Interventions: Drug: Orlistat 120 mg; Drug: Allopurinol 100 up to 600mg/day; Drug: Febuxostat 40mg Tab
- The control group (Placebo Comparator): The control group received placebo matching orlistat (tid) + standard ULT (e.g., febuxostat 40mg qd) + basic lifestyle advice (low-purine diet and exercise guidance).
  Interventions: Drug: Allopurinol 100 up to 600mg/day; Drug: Febuxostat 40mg Tab

INTERVENTIONS:
Drug: Orlistat 120 mg — Oral capsule, taken after meals, 120 mg three times daily (tid) for 24 weeks.
  Other Names: Orlistat 120 mg tid
  Arms: the experimental Group
Drug: Allopurinol 100 up to 600mg/day — Standard urate-lowering therapy (e.g., allopurinol or febuxostat), with doses adjusted based on serum uric acid levels and liver/kidney function.
Drug: Febuxostat 40mg Tab — Standard urate-lowering therapy (e.g., allopurinol or febuxostat), with doses adjusted based on serum uric acid levels and liver/kidney function.

SUMMARY:
A total of 120 obese gout patients were included in a 24-week double-blind randomized controlled design. The intervention group received orlistat 120 mg tid + UTL + individualized diet-exercise-behavioral reinforcement weight loss program, while the control group received a placebo + UTL + standard recommendations. The primary endpoint was the rate of achieving serum uric acid levels <360 μmol/L at 24 weeks; secondary endpoints included the proportion of weight loss ≥5%, frequency of gout attacks, and inflammatory indicators such as CRP and IL-1β; the activity of AMPK in PBMCs and the expression of HIF1α and NLRP3 inflammasome-related proteins were also assessed.

DETAILED DESCRIPTION:
This study employs a double-blind, randomized, controlled trial design. A total of 120 obese gout patients were included and randomly divided into two groups: the intervention group (60 cases): Orlistat (120 mg tid) + UTL + personalized dietary guidance, exercise prescription, and behavioral intervention for a duration of 24 weeks. The control group (60 cases): placebo + UTL + standard weight control recommendations, with the same intervention duration. Both groups received standard uric acid-lowering therapy (such as allopurinol or febuxostat) according to guidelines, with dosages adjusted based on blood uric acid levels and liver and kidney function to maintain stability.

Study Flow and Assessment Indicators Baseline Assessment: demographic data, medical history collection; physical examination (weight, BMI, waist circumference, etc.); laboratory tests (blood routine, urine routine, sedimentation rate, CRP, blood glucose, blood lipids, blood uric acid, liver and kidney function, etc.); collection of peripheral blood mononuclear cells (PBMCs) for mechanistic studies.

Follow-up Assessments (weeks 4, 12, 24): Clinical Indicators: changes in weight, liver and kidney function, blood lipid levels, blood uric acid levels, frequency of gout attacks.

Safety Indicators: recording of adverse events. Mechanistic Study Indicators: detection of AMPK activity in PBMCs, expression levels of HIF1α, NLRP3, ASC, caspase-1, IL-1β, and metabolomics analysis.

Statistics : SPSS 23.0; t-test/Mann-Whitney U for continuous variables, chi-square for categorical data.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the 2015 ACR/EULAR classification criteria for gout.
2. Age 18-70 years.
3. BMI ≥28 kg/m².
4. Serum uric acid ≥480 μmol/L.
5. Willing and able to comply with the study protocol.

Exclusion Criteria:

1. Contraindications to orlistat or other gout medications.
2. Severe hepatic or renal dysfunction.
3. History of severe allergy or adverse reactions to study drugs.
4. Pregnant or lactating women.
5. Malignancy.
6. Secondary gout.
7. Poor compliance or inability to cooperate.
8. Participation in other clinical trials within the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-11-09 (Estimated); Study Completion 2027-11-09 (Estimated)

PRIMARY OUTCOMES:
The rate of patients achieving target serum uric acid levels | 24 weeks
  The rate of patients achieving serum uric acid < 360 μmol/L

SECONDARY OUTCOMES:
changes in body weight | 24 weeks
  The proportion of patients with a weight loss of ≥5%,the unit of weight is Kilogram(Kg).
inflammatory markers | 24 weeks
  changes in the frequency of gout attacks, changes in inflammatory markers (CRP, IL-1β, etc.).The unit of CRP is mg/L,the unit of ESR is mm/h,the unit of IL- 1β is pg/mL.
the expression of AMPK-HIF1-inflammasome | 24 weeks
  changes in the expression of key molecules in the AMPK-HIF1-inflammasome axis.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, PLA, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] China Obesity Research Collaborative Group.Standardized Reporting for Combined Intervention Studies in Metabolic Diseases (2024 Edition)
- [Background] Chinese Rheumatology Association, Chinese Medical Association.Ethical Requirements for Clinical Trial Registration in Gout Diagnosis and Treatment Guidelines (2025 Edition)
- [Background] Chinese Evidence-Based Medicine Center, West China Hospital, Sichuan University.Operational Guidelines for Chinese Clinical Trial Registry (2023 Edition)
- [Result] Beutel ME, Dippel A, Szczepanski M, Thiede R, Wiltink J. Mid-term effectiveness of behavioral and psychodynamic inpatient treatments of severe obesity based on a randomized study. Psychother Psychosom. 2006;75(6):337-45. doi: 10.1159/000095439. PMID 17053334
- [Result] Liu S, Lin X, Tao M, Chen Q, Sun H, Han Y, Yang S, Gao Y, Qu S, Chen H. Efficacy and safety of orlistat in male patients with overweight/obesity and hyperuricemia: results of a randomized, double-blind, placebo-controlled trial. Lipids Health Dis. 2024 Mar 11;23(1):77. doi: 10.1186/s12944-024-02047-7. PMID 38468241
- [Result] Yip ASY, Leong S, Teo YH, Teo YN, Syn NLX, See RM, Wee CF, Chong EY, Lee CH, Chan MY, Yeo TC, Wong RCC, Chai P, Sia CH. Effect of sodium-glucose cotransporter-2 (SGLT2) inhibitors on serum urate levels in patients with and without diabetes: a systematic review and meta-regression of 43 randomized controlled trials. Ther Adv Chronic Dis. 2022 Mar 23;13:20406223221083509. doi: 10.1177/20406223221083509. eCollection 2022. PMID 35342538
- [Result] Sridharan K, Alkhidir MMOH. Hypouricemic effect of sodium glucose transporter-2 inhibitors: a network meta-analysis and meta-regression of randomized clinical trials. Expert Rev Endocrinol Metab. 2025 Mar;20(2):139-146. doi: 10.1080/17446651.2025.2456504. Epub 2025 Jan 21. PMID 39835962
- [Result] Chen X, Chen S, Ren Q, Niu S, Pan X, Yue L, Li Z, Zhu R, Jia Z, Chen X, Zhen R, Ban J. Metabolomics Provides Insights into Renoprotective Effects of Semaglutide in Obese Mice. Drug Des Devel Ther. 2022 Nov 9;16:3893-3913. doi: 10.2147/DDDT.S383537. eCollection 2022. PMID 36388084
- [Result] Chinese Society of Endocrinology. Guidelines for long-term weight management and clinical application of drugs in obese patients (2024 edition). Chin J Endocrinol Metab. 2024;40(7):545-564. doi:10.3760/cma.j.cn311282-20240412-00149
- [Result] Yokose C, McCormick N, Choi HK. The role of diet in hyperuricemia and gout. Curr Opin Rheumatol. 2021 Mar 1;33(2):135-144. doi: 10.1097/BOR.0000000000000779. PMID 33399399
- [Result] Larsson SC, Burgess S, Michaelsson K. Genetic association between adiposity and gout: a Mendelian randomization study. Rheumatology (Oxford). 2018 Dec 1;57(12):2145-2148. doi: 10.1093/rheumatology/key229. PMID 30085130
- [Result] Guo G, Dong C, Yin R, Yang Y, Zhao R, Wang Y, Guo J, Zhou W, Lu G. Serum urate goal attainment and associated factors in Chinese gout patients. Psychol Health Med. 2020 Sep;25(8):931-939. doi: 10.1080/13548506.2019.1706751. Epub 2019 Dec 23. PMID 31870173
- [Result] Do H, Choi HJ, Choi B, Son CN, Kim SH, Choi SR, Kim JH, Kim MJ, Shin K, Kim HO, Song R, Lee SW, Ahn JK, Lee SG, Lee CH, Son KM, Moon KW. Factors for achieving target serum uric acid levels after initiating urate-lowering therapy in patients with gout: results from the ULTRA registry. Sci Rep. 2023 Nov 22;13(1):20511. doi: 10.1038/s41598-023-47790-6. PMID 37993515
- [Result] Afinogenova Y, Danve A, Neogi T. Update on gout management: what is old and what is new. Curr Opin Rheumatol. 2022 Mar 1;34(2):118-124. doi: 10.1097/BOR.0000000000000861. PMID 34907116
- [Result] Wei J, Wang Y, Dalbeth N, Xie J, Wu J, Zeng C, Lei G, Zhang Y. Weight Loss After Receiving Anti-Obesity Medications and Gout Among Individuals With Overweight and Obese: A Population-Based Cohort Study. Arthritis Rheumatol. 2025 Mar;77(3):335-345. doi: 10.1002/art.42996. Epub 2024 Nov 11. PMID 39300602